CLINICAL TRIAL: NCT04563286
Title: Patient-Reported Outcome Measures in Wild-Type and Variant Cardiac Transthyretin Amyloidosis: The Impact of Transthyretin Amyloidosis on Life qualitY (ITALY) Study
Brief Title: Patient-Reported Outcome Measures in Wild-Type and Variant Cardiac Transthyretin Amyloidosis
Acronym: ITALY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Messina (Other)
Collaborators: Fondazione Toscana Gabriele Monasterio (Other); University of Pavia (Other); Università degli Studi di Ferrara (Other); Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Di Bella, Professor, University of Messina
Other Study IDs: IT08012020
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Transthyretin Amyloidosis
Keywords: amyloidosis; transthyretin; quality of life; score; cardiomyopathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire on life quality — Two sets of 30 PROMs questions will be created. The v-ATTR and wt-ATTR questionnaires will be critically evaluated by the whole panel, taking into account observations and feedback from patients. The 2 scores will be administered to consecutive patients evaluated at dedicated ambulatory clinics of the 4 Institutions. To confirm score reliability and responsiveness, 2 distinct patient cohorts will be recruited. The reliability cohort will be assembled to demonstrate the instrument's test-retest reliability. A second cohort of patients (responsiveness cohort) will be assembled to demonstrate the instrument's responsiveness to changes in clinical status. Patients experiencing a heart failure hospitalization within 6 months will enter the responsiveness cohort at the time of hospital admission.

SUMMARY:
Specific, standardized, comprehensive, universally accepted Patient-Reported Outcome Measures (PROMs) are currently lacking for variant and wild-type cardiac amyloid transthyretin amyloidosis (v-ATTR/wt-ATTR). Our goal is then to create two scores able to provide a cumulative assessment of cardiac involvement, peripheral neuropathy (in v-ATTR), and comorbidities, and their impact on the quality of life.

In the setting of a nationwide collaboration involving 5 main Italian referral centers for this condition (in Ferrara, Florence, Pavia, Pisa and Messina), a panel will be created, including experts of ATTR cardiomyopathy, neurologists, geriatricians, health management specialists, as well as patients with either variant or wild-type ATTR cardiomyopathy (n=50).

The most clinically relevant domains for patients (such as physical limitations, symptoms, self-efficacy and knowledge, social interference, quality of life, age-related issues, social and family environment, frailty, comorbidities) will be identified. Two sets of 30 items (one for variant and another for wild-type ATTR cardiomyopathy) will be created in collaboration with patients. Questions will be formatted for gender neutrality, clarity, interpretability, and possible foreign language translations. PROMs scores will be validated through administration to around 250 consecutive outpatients. Score performance will be evaluated in terms of internal consistency, response to clinical changes, comparison with conventional clinical measures. The time needed for completion, the clarity of questions and the need for assistance from a family caregiver will be evaluated.

This project will hopefully lead to the identification of disease-specific metrics that may serve as a clinically meaningful outcome in cardiovascular research, patient management, and quality assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cardiomyopathy due to ATTR amyloidosis, diagnosed by endomyocardial biopsy or on the basis of the algorithm for the non-invasive diagnosis of cardiac ATTR amyloidosis (Gillmore et al., 2016).
* Clinical stability, defined as the lack of unscheduled hospitalizations and/or significant changes in cardiac therapies from at least 1 month.

Exclusion Criteria:

* Lack of informed consent.
* Inability of understanding a written text in Italian.
* Absence of the conditions of clinical stability, as defined above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiac ATTR amyloidosis, either biopsy proven or diagnosed according to the algorithm for nonbiopsy diagnosis of ATTR cardiomyopathy (Gillmore et al., 2016), will be evaluated.
  PROMs for v-ATTR and wt-ATTR will be created in close collaboration with 50 patients suffering from ATTR cardiomyopathy (see below), and will be validated on a cohort of 250 patients (i.e., 50 patients from each participating center; see below).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-02-22 (Actual); Primary Completion 2022-04-22 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
reliability | baseline to 6 months
  internal consistency

SECONDARY OUTCOMES:
responsiveness | baseline to HF hospitalization (<6 months)
  changes in scores in response to clinical changes
validity of each domain | baseline to 6 months
  comparison of scores with other measures that quantify similar concepts, namely other score points, NYHA class, 6MWD, or objective measures of cardiac dysfunction, i.e. circulating levels of NT-proBNP and hs-TnT)

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Università di Ferrara, Ferrara
  - Careggi Hospital, Florence
  - Università di Messina, Messina
  - Università di Pavia, Pavia
  - Fondazione Toscana Gabriele Monasterio (FTGM), Pisa

IPD SHARING:
Plan to Share IPD: Undecided